CLINICAL TRIAL: NCT04409938
Title: The Effect of Progressive Muscle Relaxation and Nature Sounds on Blood Pressure Measurement Skills, Anxiety Levels, and Vital Signs in Nursing Students
Brief Title: Progressive Muscle Relaxation and Nature Sounds in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevda Korkut, Principal Inverstigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 121
Record Dates: First submitted 2020-05-21; First posted 2020-06-01 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Anxiety
Keywords: Skill training; Nursing students; Anxiety; Blood Pressure Measurement Skills
MeSH Terms: conditions — Anxiety Disorders | interventions — Autogenic Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive Muscle Relaxation (Experimental): PMR participants rested for ten minutes between the sessions and then practiced PMR for 15 minutes. PMR consisted of taking a deep breath five times and then clenching fists, raising the shoulders, bringing the forearms towards the body, stretching the triceps muscle, and tensing and relaxing the forehead, eye, chin, neck, chest, abdomen, back, hips, thigh, and feet muscles. The investigators made a video of exercises in a certain order and uploaded it to the television in the lab prior to the intervention.
  Interventions: Other: Progressive Muscle Relaxation
- Progressive Muscle Relaxation with Nature Sounds (Experimental): PMR+NS participants practiced PMR accompanied by nature sounds.
  Interventions: Other: Progressive Muscle Relaxation; Other: Nature Sounds
- Standard Practice (No Intervention): The standard practice of the lab was made.

INTERVENTIONS:
Other: Progressive Muscle Relaxation — PMR participants rested for ten minutes between the sessions and then practiced PMR for 15 minutes. PMR consisted of taking a deep breath five times and then clenching fists, raising the shoulders, bringing the forearms towards the body, stretching the triceps muscle, and tensing and relaxing the forehead, eye, chin, neck, chest, abdomen, back, hips, thigh, and feet muscles. The investigators made a video of exercises in a certain order and uploaded it to the television in the lab prior to the intervention. The investigators turned on the video during the intervention and asked the participants to follow the instructions for PMR exercises.
  Arms: Progressive Muscle Relaxation; Progressive Muscle Relaxation with Nature Sounds
Other: Nature Sounds — PMR+NS participants practiced PMR accompanied by nature sounds. PMR consisted of taking a deep breath five times and then clenching fists, raising the shoulders, bringing the forearms towards the body, stretching the triceps muscle, and tensing and relaxing the forehead, eye, chin, neck, chest, abdomen, back, hips, thigh, and feet muscles. The investigators made a video of exercises in a certain order and uploaded it to the television in the lab prior to the intervention. The investigators turned on the video during the intervention and asked the participants to follow the instructions for PMR exercises.
  Arms: Progressive Muscle Relaxation with Nature Sounds

SUMMARY:
Background: The aim of this study was to determine the effect of PMR and nature sounds on nursing students' BPM skills, and anxiety levels and vital signs.

Methods: This was a randomized controlled experimental study conducted at the nursing department of the faculty of health sciences of a university. PMR participants rested for ten minutes between the sessions and then practiced PMR for 15 minutes. PMR+NS participants practiced PMR accompanied by nature sounds.

DETAILED DESCRIPTION:
Background: The aim of this study was to determine the effect of PMR and nature sounds on nursing students' BPM skills, and anxiety levels and vital signs.

Methods: This was a randomized controlled experimental study conducted at the nursing department of the faculty of health sciences of a university. PMR participants rested for ten minutes between the sessions and then practiced PMR for 15 minutes. PMR consisted of taking a deep breath five times and then clenching fists, raising the shoulders, bringing the forearms towards the body, stretching the triceps muscle, and tensing and relaxing the forehead, eye, chin, neck, chest, abdomen, back, hips, thigh, and feet muscles. The investigators made a video of exercises in a certain order and uploaded it to the television in the lab prior to the intervention. The investigators turned on the video during the intervention and asked the participants to follow the instructions for PMR exercises. PMR+NS participants practiced PMR accompanied by nature sounds.

ELIGIBILITY:
Inclusion Criteria:

1. being a first-year nursing student
2. voluntary
3. participating in the theoretical part of the "Pulse and Blood Pressure Measurement" course and in lab practice.

Exclusion Criteria:

* not participating in the theoretical part of the "Pulse and Blood Pressure Measurement" course and in lab practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAI) | pre-intervention
  The STAI consists of two parts; the State Anxiety Inventory (SAI) and the Trait Anxiety Inventory (TAI). The SAI measures anxiety about an event while the TAI measures anxiety level as a personal characteristic. The TAI and SAI each consists of 20 items. The SAI items are scored on a 4-point Likert scale of 1 to 4 (1= never, 2= sometimes, 3= often, 4= always). The SAI items are scored on a 4-point Likert scale of 1 to 4 (1= almost never, 2= sometimes, 3= often, 4= almost always). Ten SAI items (1, 2, 5, 8, 10, 11, 15, 16, 19, and 20) and six TAI items (1, 6, 7, 13, 16, and 19) are reverse scored. Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
The State Anxiety Inventory (SAI) | through study completion for each group, an average of 4 hour
  The SAI items are scored on a 4-point Likert scale of 1 to 4 (1= almost never, 2= sometimes, 3= often, 4= almost always). Ten SAI items (1, 2, 5, 8, 10, 11, 15, 16, 19, and 20) and six TAI items (1, 6, 7, 13, 16, and 19) are reverse scored. Higher scores indicate greater anxiety
The Blood Pressure Knowledge Test (BPKT) | through study completion for each group, an average of 4 hour
  BPKT is a multiple-choice test consisting of 20 items on definitions, physiology, affecting factors, classification, measurement sites, planning, application auscultation/ palpation measurement, and evaluation. A correct response is scored 1, and therefore, the total score ranges from 0 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda Korkut, PhD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)